CLINICAL TRIAL: NCT00592644
Title: Laser Atraumatic Treatment Of Ectasias On Vocal Cords
Brief Title: Laser Treatment Of Vascular Lesions On Vocal Cords
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Zhi Wang, Trustees of Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDC-006853A; R21DC006853 (NIH); R21-006853-2
Record Dates: First submitted 2007-12-31; First posted 2008-01-14 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Ectasia
Keywords: ectasia; vascular lesions; vocal cords; voice; pulsed dye laser
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Fibrillins; Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pulse Dye Laser
  Interventions: Procedure: Pulse Dye laser (PDL)
- 2 (Active Comparator): Traditional surgeries
  Interventions: Procedure: CO2 laser or other traditional surgeries

INTERVENTIONS:
Procedure: Pulse Dye laser (PDL) — one-time PDL, in 10 subjects
  Other Names: the laser made by Cynosure Inc, Mass
  Arms: 1
Procedure: CO2 laser or other traditional surgeries — once-time CO2 laser or other conventional surgeries, in other 10 subjects
  Other Names: the laser made by Cynosure Inc. Mass
  Arms: 2

SUMMARY:
Small vascular malformations (SVM) on the vocal fold is a common problem that can disturb the voice. The pulsed dye laser (PDL) has been successfully used for treatment of blood vessel abnormalities in surface tissue, through its high selectivity for destroying targeted blood vessels while sparing normal tissue. However, there is no study to determine its clinical benefit for treatment of SVMs on vocal fords. In this proposed study, we plan to make such a determination.We will determine whether PDL will produce better and quicker voice improvement than the conventional surgeries, in 20 patients (10 cases of each group) with vocal fold SVM. We expect that this less invasive laser treatment will provide an ideal and excellent option for this disease.

DETAILED DESCRIPTION:
Clinically, small vascular malformations (SVM) on the vocal fold is a common problem that can disturb the voice. Currently, this problem is treated with endoscopic microsurgery with the use of a Carbon dioxide (CO2) laser or other microsurgeries. However, those treatments are unsatisfactory because of their invasive nature. The pulsed dye laser (PDL) has been successfully used for treatment of blood vessel abnormalities in surface tissue, through its high selectivity for destroying targeted blood vessels while sparing normal tissue. Even thought this process has been in use clinically for the past 5 years, there is no study to determine its clinical benefit for treatment of SVMs on vocal fords, by comparing it with routine surgeries. In this proposed study, we plan to make such a determination, by comparing the voice recovery and voice improvement between this laser and those routine surgeries (with CO2 laser or "cold" instrument).

Our specific aim is to determine whether PDL will produce better and quicker voice improvement than the conventional surgeries, in 20 patients (10 cases of each group) with vocal fold SVM. This is the first study to determine clinical benefit of the microvascular targeting (MVT) technique of laser to treat vocal fold SVMs, by a comparison of the voice results between these two groups. We expect that this less invasive laser treatment will provide an ideal and excellent alternative to current surgical approaches for treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. have SVMs or other small (2.0 mm diameter or less) vasculature-related lesions on vocal fold
2. Hoarseness or other symptoms of alteration in phonation is persistent least for 3 months
3. have (or have a high risk of) recurrent vocal fold hemorrhage, SVM enlargement or persistent fold vibratory abnormality
4. 18 years of age or older
5. Failure to response to voice training or other non-surgical treatments
6. Require CO2 laser ablation or other surgical removal of the lesion
7. Willingness to participate in a 6-month study and adhere to the follow-up schedule
8. A signed informed consent form

Exclusion Criteria:

1. Age less than 18 years, or older than 64
2. Any evidence of mental impairment such that the patient cannot understand the protocol or be in a position to sign the informed consent form
3. Clinical or histological evidence of malignant conversion
4. Lesion to be larger than 2.00 mm diameter or those non-vascular lesions
5. Pregnant women
6. Severity of disease such that airway patency is in immediate danger
7. Patients for whom the voice quality is particularly important: including signers, actors, or other similar professions or person who requires a very high voice quality

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2005-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Recovery of Voice | 5 months

SECONDARY OUTCOMES:
clearance of lesion | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Wang, MD, Principal Investigator — Boston University